CLINICAL TRIAL: NCT02713282
Title: A 52-Week, Open-Label, Prospective, Multicenter, International Study of a Transition to the Paliperidone Palmitate 3-Month Formulation In Patients With Schizophrenia Previously Stabilized on the Paliperidone Palmitate 1-Month Formulation
Brief Title: A Study of Transition to the Paliperidone Palmitate 3-Month Formulation In Participants With Schizophrenia Previously Stabilized on the Paliperidone Palmitate 1-Month Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108121; 2015-004835-10 (EudraCT Number); R092670SCH3015 (Other: Janssen-Cilag Limited); NCT02772393 (obsolete NCT alias)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; R092670; Paliperidone Palmitate
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Paliperidone palmitate 3 month formulation (PP3M) (Experimental): Participants will receive intramuscular injection of Paliperidone Palmitate 3-Month Formulation (PP3M) on Day 1 at a starting dose of 175 milligram equivalent (mg eq.) up to 525 mg eq. based on last Paliperidone Palmitate 1-Month Formulation (PP1M) dose (at a dose of 3.5-fold multiple of the participant's last PP1M dose). Subsequent PP3M injections will be given at Month 3, Month 6, and Month 9 and dose can be adjusted flexibly in increments within the range of 175 to 525 mg eq.
  Interventions: Drug: Paliperidone palmitate 3 month formulation (PP3M)

INTERVENTIONS:
Drug: Paliperidone palmitate 3 month formulation (PP3M) — Participants will receive intramuscular injection of Paliperidone Palmitate 3-Month Formulation (PP3M) on Day 1 at a starting dose of 175 milligram equivalent (mg eq) up to 525 mg eq based on last Paliperidone Palmitate 1-Month Formulation (PP1M) dose (at a dose of 3.5-fold multiple of the participant's last PP1M dose). Subsequent PP3M injections will be given at Month 3, Month 6, and Month 9 and dose can be adjusted flexibly in increments within the range of 175 to 525 mg eq.

SUMMARY:
The purpose of this study is to estimate the proportion of participants fulfilling criteria for symptomatic remission following a transition to 12 months treatment with flexible-dose paliperidone palmitate 3 month formulation (PP3M) in participants with schizophrenia previously adequately treated with paliperidone palmitate 1 month formulation (PP1M) for at least 4 months.

DETAILED DESCRIPTION:
This is an international, multicenter (study conducted at multiple sites) study designed to estimate remission rates and assess treatment response, tolerability, and patterns of use of Paliperidone Palmitate 3-Month Formulation (PP3M) in a diverse population of participants with schizophrenia. The study will consist of a screening phase (Day -7 to Day 1), a 52-week, open-label, flexible-dose PP3M treatment phase and a follow up safety assessment 3 months ( +/-14 days ) after the month 12 visit or early discontinuation. Participants' Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria for a diagnosis of schizophrenia
* Able to read, understand, and sign the informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study
* Willing and able to fill out self-administered questionnaires
* Willing and able to adhere to the prohibitions and restrictions specified in the protocol
* A woman of childbearing potential must have a negative urine pregnancy test at Screening and baseline
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study drug

Exclusion Criteria:

* His/her psychiatric diagnosis is due to direct pharmacological effects of a substance (example, a drug of abuse or medication) or a general medical condition (example, clinically notable hypothyroidism, organic brain disorder)
* Experienced intolerable side effects during treatment with paliperidone palmitate 1-month formulation (PP1M)
* Has a known hypersensitivity to paliperidone or risperidone
* Has received any other long-acting injectable antipsychotic medication other than PP1M within the last 4 months before the first injection of the study drug paliperidone palmitate 3-month formulation (PP3M)
* Has received clozapine during the last 3 months before the Screening visit
* Is considered to be at imminent risk of suicide, even after clinical intervention
* Has a serious unstable medical condition, including recent and present clinically relevant laboratory abnormalities
* Has a history or current symptoms of tardive dyskinesia or neuroleptic malignant syndrome
* Is a woman who is pregnant or breast-feeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of PP3M
* Has participated in an investigational drug trial in the 30 days prior to the Screening visit or is currently enrolled in an investigational study
* Has a current DSM-5 diagnosis of dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, autistic disorder, or intellectual disabilities and/or meets the DSM-5 definition of severe substance use disorder (except for nicotine and caffeine) within 6 months prior to screening; however, participants with mild or moderate substance use disorder, with the exception of intravenous drug use, will be eligible for enrollment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Symptomatic Remission Based on Positive and Negative Syndrome Scale (PANSS) | Month 12
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent), 2 (minimal), 3 (mild), 4 (moderate), 5 (moderately severe), 6 (severe) and 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity. Symptomatic remission is defined as achieving intensity level of mild or moderate on PANSS scale by all 8 items as the determinants for symptomatic remission: delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/posturing, blunted affect, social withdrawal, lack of spontaneity.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Symptomatic Remission Based on Positive and Negative Syndrome Scale (PANSS) at Month 6, 9 and 12 | Month 6, Month 9 , and Month 12
  PANSS is a 30-item scale to assess neuropsychiatric symptoms of schizophrenia. PANSS provides a total score and scores for 3 subscales, positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items), each item scored on a scale of 1 (absent), 2 (minimal), 3 (mild), 4 (moderate), 5 (moderately severe), 6 (severe) and 7 (extreme). Total score ranges from 30 to 210 and higher score indicates greater severity. Symptomatic remission is defined as achieving intensity level of mild or moderate on PANSS scale by all 8 items as the determinants for symptomatic remission: delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/posturing, blunted affect, social withdrawal, lack of spontaneity with the achieved intensity level maintained for at least 6 months.
Time to Symptomatic Remission | Up to Month 12
  Time to Symptomatic Remission will be reported. Symptomatic remission is defined as achieving intensity level of mild or moderate on PANSS scale by all 8 items as the determinants for symptomatic remission: delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/posturing, blunted affect, social withdrawal, lack of spontaneity with the achieved intensity level maintained for at least 6 months.
Percentage of Participants who Meet the Remission Severity Criteria | Up to Month 12
  Remission severity criteria that is, a score of mild or less [less than or equal to 3] on all selected PANSS items [P1, P2, P3, N1, N4, N6, G5, and G9]) at each time point.
Non-Inferiority of Change in PANSS Total Score From Baseline to Month 12 last-observation-carried-forward (LOCF) | Up to Month 12
  Maintained efficacy will be investigated using the Schuirmann's test to test the change at last-observation-carried-forward (LOCF) endpoint in total PANSS score at endpoint versus baseline with a non-inferiority margin of 5 points on the PANSS scale.
The proportion of subjects with PANSS response | Up to Month 12
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent), 2 (minimal), 3 (mild), 4 (moderate), 5 (moderately severe), 6 (severe) and 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Limited Clinical Trial, Study Director — Janssen-Cilag Limited
Locations (46):
- Croatia (2):
  - Rijeka
  - Zagreb
- Esbjerg, Denmark
- France (5):
  - Clermont-Ferrand
  - Montpellier
  - Paris
  - Rennes
  - Toulon
- Germany (4):
  - Berlin
  - Hamburg
  - Oranienburg
  - Stralsund
- Greece (4):
  - Athens
  - Heraklion
  - Nea Kifissia
  - Thessaloniki
- Israel (2):
  - Beer Yaakov
  - Ramat Gan
- Malaysia (3):
  - Ipoh
  - Johor Bahru
  - Kuala Lumpur
- Netherlands (2):
  - Assen
  - Groningen
- Russia (2):
  - Moscow
  - Saint Petersburg
- Jeddah, Saudi Arabia
- South Korea (4):
  - Gwangju
  - Gyeonggi-do
  - Jeonju
  - Seoul
- Spain (6):
  - Bilbao
  - Madrid
  - Oviedo
  - Sabadell
  - Torrevieja
  - Valencia
- Taiwan (3):
  - New Taipei City
  - Tainan
  - Taoyuan District
- Turkey (Türkiye) (4):
  - Ankara
  - Bursa
  - Istanbul
  - Sakarya
- United Kingdom (3):
  - Derby
  - Edinburgh
  - Reading

REFERENCES:
- [Derived] Pungor K, Bozikas VP, Emsley R, Llorca PM, Gopal S, Mathews M, Wooller A, Bergmans P. Stable patients with schizophrenia switched to paliperidone palmitate 3-monthly formulation in a naturalistic setting: impact of patient age and disease duration on outcomes. Ther Adv Psychopharmacol. 2020 Dec 23;10:2045125320981500. doi: 10.1177/2045125320981500. eCollection 2020. PMID 35186258
- See also: Related Info — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-004835-10/results